CLINICAL TRIAL: NCT02054195
Title: Study of Special Guided Training Model on Insertion Techniques for Postplacental Intra Uterine Device to Prevent Expulsion
Brief Title: Training Model on Insertion Techniques for Postplacental Intra Uterine Device
Acronym: PTKP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Showa University (Other)
Responsible Party: Principal Investigator, Yuditiya Purwosunu, MD, Showa University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: jm1
Record Dates: First submitted 2014-01-25; First posted 2014-02-04 (Estimated); Last update posted 2014-02-04 (Estimated); Status verified 2014-02

CONDITIONS: Intra-uterine Device Complication

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- IUD new technique (Experimental): Training
  Interventions: Behavioral: Training
- No Training (Experimental): No Training
  Interventions: Behavioral: No Training

INTERVENTIONS:
Behavioral: Training — Training model is consist of effort to provide intra uterine device post placental by organising a special guided training model for post-placental IUD insertion by pushing the head of IUD using index and middle finger close enough to fundal part of uterus to prevent expulsion.
  Arms: IUD new technique
Behavioral: No Training — Control of Training model is without training on effort of pushing the head of IUD using index and middle finger to uterine fundus.
  Arms: No Training

SUMMARY:
This study aimed to compare special guided training model with standard procedure on insertion technique for post-placental intra uterine device that provides IUD location close enough to fundal part of uterus to prevent expulsion

DETAILED DESCRIPTION:
The standard of insertion IUD postplacental can not provide prevention of expulsion. Special techniques on insertion IUD is needed for preventing expulsion. This training model is consisted of the special techniques to provide intra uterine device post placental close enough to fundal part of uterus to prevent expulsion

ELIGIBILITY:
Inclusion Criteria:

* 37-42 weeks gestation pregnancy women in delivery, singleton pregnancy, without any uterine anomaly

Exclusion Criteria:

* Any bleeding and infection complication

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 230 (Actual)
Dates: Start 2012-08; Primary Completion 2013-09 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Number of Participants with IUD total or partial expulsion | 12 Months
  Transabdominal ultrasonography examination was done by researcher right after insertion. Ultrasonography examination was done using longitudinal and transversal scan, with client in supine position using real time convex 2 probe with 3,5 Mhz frequency. While transvaginal ultrasonography examination was done when the client come after 6 weeks, 6 months and 12 months after insertion.

SECONDARY OUTCOMES:
Percentage of Participants with retained skill and knowledge | 12 Months

CONTACTS AND LOCATIONS:
Overall Officials: Seno Adjie, MD, PhD, Principal Investigator — Indonesia University
Locations (1):
- Central nationalHospital Cipto Mangunkusumo, Jakarta, Jakarta Special Capital Region, Indonesia